CLINICAL TRIAL: NCT05139186
Title: The EYE Study: Enhancing the Diagnostic Yield of Standard Colonoscopy by Artificial Intelligence Aided Endoscopy
Brief Title: The EYE Study Enhancing the Diagnostic Yield of Standard Colonoscopy by Artificial Intelligence Aided Endoscopy
Acronym: EYE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 3000
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Artificial Intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WL+AI (Experimental): Colonoscopy in white light and artificial intelligence
  Interventions: Device: Artificial Intelligence
- WL (Experimental): Colonoscopy in white light
  Interventions: Device: Artificial Intelligence

INTERVENTIONS:
Device: Artificial Intelligence — Artificial intelligence

SUMMARY:
Colorectal cancer (CRC) remains one of the leading causes of mortality among neoplastic diseases in the world[1] . Adequate colonoscopy based CRC screening programs have proved to be the key to reduce the risk of mortality, by early diagnosis of existing CRC and detection of pre-cancerous lesions[2-4] . Nevertheless, long-term effectiveness of colonoscopy is influenced by a range of variables that make it far from a perfect tool[5]. The effectiveness of a colonoscopy mainly depends on its quality, which in turn is dependent on the skill and expertise of the endoscopist. In fact, several studies have shown a significant adenoma miss rate of 24%-35%, especially in patients with diminutive adenomas[6,7] . These data are in line with interval cancers incidence (I-CRC), defined as the percentage of cancers diagnosed after a screening program and before the intended surveillance duration, of approximately 3%-5% [8,9].

The development of the artificial intelligence (AI) applications in the medical field has grown in interest in the past decade. Its performance on increasing automatic polyp and adenoma detection has shown promising results in order to achieve an higher ADR[10]. The use of computer aided diagnosis (CAD) for detection of polyps had initially been studied in ex vivo studies but in the last few years, with the advancement in computer aided technology and emergence of deep learning algorithms, use of AI during colonoscopy has been achieved and more studies have been undertaken [10].

Recently Fujifilm (Tokyo, Japan) has developed a new technology known as "CAD-EYE" aiming to support both colonic polyp detection and characterization during colonoscopy. This technology is now available in Europe, being compatible with the latest generation of Fujifilm endoscopes (ELUXEO Fujifilm Co.).

However, the clinical impact of CAD-EYE system in improving the adenoma detection have yet to be assessed

ELIGIBILITY:
Inclusion Criteria:

- patients aged 45 or older undergoing average risk colonoscopy (screening) or follow-up colonoscopy for previous history of polyps (surveillance interval of 3 years or greater).

Exclusion Criteria:

* subjects with personal history of CRC, or IBD.
* subjects affected with Lynch syndrome or Familiar Adenomatous Polyposis.
* patients with inadequate bowel preparation (defined as Boston Bowel Preparation Scale < 2 in any colonic segment).
* patients with previous colonic resection.
* patients on antithrombotic therapy, precluding polyp resection.
* patients who were not able or refused to give informed written consent.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1120 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Adenoma per colonoscopy (APC) | 9 Months
  APC, defined as the total number of histologically confirmed adenomas and carcinomas detected in the colonoscopy divided by the total number of colonoscopies.

SECONDARY OUTCOMES:
Positive predictive value (PPV) | 9 Months
  PPV, defined as the total number of histologically confirmed adenomas and carcinomas detected during the colonoscopy, divided by the total number of excisions in the colonoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No